CLINICAL TRIAL: NCT02292628
Title: Study Phase I/II, Double Blind, Randomized, Comparing Two Groups to Evaluate the Safety and Efficacy of Autologous Mesenchymal Stem Cells From Adipose Tissue (CMMAd) in the Treatment of the Faecal Incontinence
Brief Title: Study, Double Blind, Randomized, Comparing Two Groups to Evaluate the Safety and Efficacy of Autologous Mesenchymal Stem Cells From Adipose Tissue (CMMAd) in the Treatment of the Faecal Incontinence
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Andalusian Initiative for Advanced Therapies - Fundación Pública Andaluza Progreso y Salud (Other)
Collaborators: Iniciativa Andaluza en Terapias Avanzadas (Other)
Responsible Party: Sponsor
Organization: Andalusian Network for Design and Translation of Advanced Therapies (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CMMAd/InFe/2011
Record Dates: First submitted 2014-11-06; First posted 2014-11-17 (Estimated); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Faecal Incontinence
MeSH Terms: conditions — Encopresis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mesenchymal stem cells (Experimental): Autologous mesenchymal stem cells from the adipose tissue in an unique intralesional infusion with a dose of 40 million cells.
  Interventions: Drug: Infusion of mesenchymal stem cells from adipose tissue
- Ringer lactate solution (Placebo Comparator): Ringer lactate solution
  Interventions: Other: Infusion of placebo

INTERVENTIONS:
Drug: Infusion of mesenchymal stem cells from adipose tissue
  Arms: Mesenchymal stem cells
Other: Infusion of placebo
  Arms: Ringer lactate solution

SUMMARY:
This is a clinical trial phase I/II, double blind, randomized to compare in two groups of patients to evaluate the safety and efficacy of the autologous mesenchymal stem cells from the adipose tissue (CMMAd) in the treatment of the faecal incontinence.

DETAILED DESCRIPTION:
In the phase of recruitment, of 20 months of duration, there will be included 16 participants who will be randomized to one of the groups of intervention (8 patients group CMMAd / 8 patients group placebo). The phase of follow-up of every patient will be 12 months, though, provided that these patients are seen regularly in the study sites of the study, once concluded his follow-up will be continued to be able to obtain safety information and efficacy to 24 months.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females in the age group of 18-80 yrs.
2. A unique internal sphincter defect and / or external (no more than 100 º), at any level of the anal canal, of any cause (except those described in the exclusion criteria).
3. Severity of faecal incontinence of 12 or more in the Wexner Score and / or at least six episodes of faecal incontinence for a period of 28 days.
4. Duration of faecal incontinence of at least two years prior to inclusion.
5. Patients who are able to understand the requirements of the study, and willing to provide voluntary written informed consent.

Exclusion Criteria:

1. More of an external sphincter defect and / or at any level of internal anal canal.
2. Have received treatment to faecal failure with bulking agents, neuromodulation or surgery.
3. Current anorectal tumors.
4. Current anal fissures.
5. Anorectal stenosis
6. Chronic pelvic or anorectal pain.
7. Pregnant or 6 months postpartum.
8. Medical history of infection with Human Immunodeficiency Virus (HIV) or any severe immunocompromised state or therapy immunosuppressive.
9. Malignancies in remission for less than a year before the study. An exception to the basocellular carcinoma (BCC) in "remission" for less than a year.
10. Bleeding diathesis or current anticoagulant therapy.
11. Chemotherapy during the 6 months preceding the study.
12. Previous radiation with evidence of radiation injury in the treated area.
13. Participation in any other clinical study during the 3 months preceding the pre-study visit.
14. Patients with other serious disorders.
15. Patients with uncontrolled inflammatory disease or taking drugs prohibited in the protocol or active perianal disease.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2013-10; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Number of Serious Adverse Events | 12 months

SECONDARY OUTCOMES:
Changes in the faecal incontinence diary | 12 months
Anorectal manometry | 12 months
Jorge-Wexner Score | 12 months
Faecal Incontinence Quality of Life | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Fernando de la Portilla, Dr., Principal Investigator — Hospital U. Virgen del Rocio; Santiago Mera, Dr., Principal Investigator — Hospital Regional U de Málaga
Locations (4):
- Spain (4):
  - H. Juan Ramón Jiménez, Huelva
  - Fundación Jiménez Díaz, Madrid
  - Hospital Regional U de Málaga, Málaga
  - Hospital U Virgen del Rocio, Seville